CLINICAL TRIAL: NCT03251885
Title: Extended-spectrum β-lactamase-producing Enterobacteriaceae (ESBL) Vertical Carriage and Transmission Rates in Women With Preterm Labor Versus Women With Term Pregnancy
Brief Title: Extended-spectrum β-lactamase -Producing Enterobacteriaceae (ESBL) Vertical Transmission in Women With Preterm Labor Versus Those in Term Pregnancy
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Western Galilee Hospital-Nahariya (Other Government)
Responsible Party: Principal Investigator, Dr. Maya Wolf, MD, Western Galilee Hospital-Nahariya
Other Study IDs: 0188-16-NHR
Record Dates: First submitted 2017-08-14; First posted 2017-08-16 (Actual); Last update posted 2021-03-08 (Actual); Status verified 2021-03

CONDITIONS: Preterm Labor
MeSH Terms: conditions — Obstetric Labor, Premature

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Two swabs will be taken at each screen: one from the vagina and the other from the rectum for vaginal and rectal assessment of maternal colonization. Maternal colonizing ESBL strain will be compared with infant's strain, if detected by the routine weekly NICU rectal surveillance for ESBL carriage.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- women with preterm labor: pregnant women < 37 weeks of gestations with regular uterine contractions and > 3 cm dilation, > 80% effacement
  Interventions: Other: swabs
- women with term pregnancy: pregnant women > 37 weeks of gestation
  Interventions: Other: swabs

INTERVENTIONS:
Other: swabs — Two swabs will be taken at each screen: one from the vagina and the other from the rectum for vaginal and rectal assessment of maternal colonization

SUMMARY:
The aims of the study are to evaluate the rate of ESBL-producing Enterobacteriaceae colonization among women in preterm labor and term labor, the incidence of maternal vertical transmission of ESBL, and the clinical significance of ESBL in preterm infants.

DETAILED DESCRIPTION:
Preterm delivery occurs before 37 weeks of gestation. Worldwide the preterm birth rate is estimated to be about 11% and in Israel the preterm birth rate is approximately 7% (1, 2). Preterm birth is the leading direct cause of neonatal death (death in the first 28 days of life), and is responsible for 27% of neonatal deaths worldwide. Preterm births are divided to spontaneous, due to preterm labor or preterm premature rupture of membrane, or iatrogenic with labor induction due to maternal or fetal complications. The major risk factors for spontaneous preterm birth include previous preterm delivery, multiple gestation, uterine anomaly, systemic infection, history of cervical surgery and short cervical length. The clinical findings of true labor (contractions plus cervical changes) are the same whether labor occurs preterm or at term (3).

Treatment of women <34 weeks of gestation with suspected preterm labor consist of a course of betamethasone to reduce neonatal morbidity and mortality associated with preterm birth, tocolytic drugs for up to 48 hours to delay delivery, antibiotics for Group B Streptococcus (GBS) chemoprophylaxis and magnesium sulfate for pregnancies at 24 to 32 weeks of gestation to provide neuroprotection against cerebral palsy and other types of severe motor dysfunction (4). A 2014 Cochrane review of randomized trials of intrapartum antibiotic treatment of women colonized with GBS found that intrapartum antibiotic prophylaxis resulted in a significant reduction in early-onset neonatal GBS infection and a non-significant reduction in neonatal mortality (5). Intrapartum antibiotic prophylaxis is given in cases of positive screening culture for GBS from either vagina or rectum, positive history of birth of an infant with early-onset GBS disease or GBS bacteriuria during the current pregnancy (6, 7, 8). Other risk factors of developing early-onset sepsis include Intrapartum fever ≥38ºC, preterm labor (<37 weeks of gestation) and prolonged rupture of membranes (≥18 hours); women who have these risk factors should receive antibiotic prophylaxis in labor (9).

The Israeli Center for Disease Control report concerning early-onset neonatal invasive GBS disease showed a relatively similar incidence of invasive disease over the years 2006-2015 (10). In contrast, a recent report showed a marked increase in Gram-negative early-onset sepsis. The incidence of early-onset Gram-negative sepsis in Israel during the years 2008-2014 was 0.49 for 1000 live births and increased from 0.16 per 1000 in 2008 to 0.32 in 2014 (11). The incidence of E.coli early-neonatal sepsis rises significantly in preterm births (55 in preterm births vs. 26 in term) and in 2014 the burden of disease caused by E.coli was higher than GBS.

Most Gram-negative pathogens are resistant to ampicillin. Resistance of isolated E.coli to second and third generation cephalosporins was noted in 8.3% of early-onset infections, particularly in preterm and low-birth weight neonates and imply transmission of resistant strains during labor. Extended-spectrum β- lactamase-producing Enterobacteriaceae (ESBL) are pathogens which are practically resistant to all penicillins and cephalosporines. ESBL- producing Enterobacteriaceae may also harbor additional antibiotic-resistant genes against aminoglycosides, trimethoprim-sulfamethoxazole, ciprofloxacin and other agents (12). Although the prevalence of ESBL carriage is unknown, it is clearly increasing in the community and in many parts of the world 10-40% of strains of E.coli and Klebsiella pneumoniae express ESBL. However, there are no guidelines concerning surveillance cultures of pregnant women both in term or preterm labor for ESBL colonization although neonatal screening in neonatal intensive care units (NICU), on admission and periodically after, is accepted in order to prevent ESBL transmission in the NICU. In addition, we would like to compare the rate of ESBL carriage rate in women in preterm versus term labor.

ELIGIBILITY:
Inclusion Criteria:

* Preterm delivery <37 weeks of gestation
* term delivery > 37 weeks of gestation

Exclusion Criteria:

* Unknown gestational age

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Gender Based: Yes — female only
Study Population: women in preterm labor women in term labor
Sampling Method: Probability Sample
Enrollment: 300 (Estimated)
Dates: Start 2017-04-12 (Actual); Primary Completion 2021-12 (Estimated); Study Completion 2022-06 (Estimated)

PRIMARY OUTCOMES:
Maternal rectal and vaginal specimens will be compared to assess influence of culturing site and admission and labor specimens will be compared for possible influence of hospitalization on ESBL carriage | two years
  positive ESBL vs. negative ESBL

CONTACTS AND LOCATIONS:
Overall Officials: Maya Wolf, MD, Principal Investigator — Galilee Medical Center
Locations (1):
- Galil Medical Center, Nahariya, Israel

REFERENCES:
- [Derived] Sgayer I, Glikman D, Shqara RA, Maimon M, Rechnitzer H, Lowenstein L, Wolf MF. Maternal colonization with extended-spectrum beta-lactamase-producing Enterobacteriaceae in term versus preterm pregnancies. Int J Gynaecol Obstet. 2023 May;161(2):447-454. doi: 10.1002/ijgo.14555. Epub 2022 Nov 22. PMID 36334053